CLINICAL TRIAL: NCT04147988
Title: Describing, Detecting and Orienting Adults Without Intellectual Disability Asking for an Autism Spectrum Disorder Diagnosis
Brief Title: Characterizing ASD Adult Population Asking for a Diagnosis
Acronym: ASSORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A01130-57
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: adult patients without intellectual disability (IQ> 70 or college-level equivalent) and being on the waiting list for a diagnosis of ASD at the former Donald-T unit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DONALD T list (Other): adults on the DONALD T list seeking diagnostic advice on autism spectrum disorder or asperger's syndrome
  Interventions: Other: screening and diagnostic assessment DONALD T unit list

INTERVENTIONS:
Other: screening and diagnostic assessment DONALD T unit list — Screening and diagnostic assessment of the group of people awaiting assessment, and thus test the feasibility of a screening and diagnosis procedure for autism in adults without intellectual disabilities

SUMMARY:
The investigators aim at offering to about 80 patients a diagnostic assessment for Autism Spectrum Disorder (ASD), and at testing the feasibility of this protocol to detect and diagnose ASD in adults without intellectual disability.

DETAILED DESCRIPTION:
About 80 adults asked for an ASD diagnosis a Donald-T unit, now closed.The investigators will offer to these patients a diagnostic assessment, with questionnaires, ADOS-II, Vineland Adaptative Behavior Scale and psychiatric examination. Patients who will show negative scores at the detecting questionnaires will not be further assessed, except for 10 out of them, who will be drawn by lot. Then the investigators will be able to discuss the feasibility of such a procedure with these tools, as well as to describe the clinical profile of adult people asking for ans ASD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* to be on Donald-T's waiting list
* be at least 18 years old

Exclusion Criteria:

* Any participant who does not meet the inclusion criteria will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Autism Diagnostic Observation Schedule (ADOS-2) | 3 months
  Autism Diagnostic Observation Schedule (ADOS-2),Scale of observation for the diagnosis of autism.Interactive semi structured direct observation tool. Four modules adapted according to language and level of development. Module 4 is applicable to a teenager or adult with fluent language (consisting of desquestions and conversation).To evaluate social interactions, communication, play and imagination
Adult Asperger's Assessment (AAA) | 3 months
  Semi-structured clinical interview, with the patient and an informant, To evaluate social interaction, restricted activities, communication, magination, additional criteria

SECONDARY OUTCOMES:
Vineland Adaptative Behavior Scale (VABS-2) | 3 months
  The Vineland Adaptative Behavior Scale (VABS-2) is designed to measure adaptive behavior of individuals from birth to age 90. The Vineland-II contains 5 domains each with 2-3 subdomains. The main domains are: Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior (optional).
Hospital Anxiety and Depression Scale (HADS) | 3 months
  The Hospital Anxiety and Depression Scale (HADS) is an instrument for detecting anxiety and depressive disorders. It has 14 listed items from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), allowing thus obtaining two scores (maximum score of each score = 21).
Liebowitz Social Anxiety Scale (LSAS) | 3 months
  The Liebowitz Social Anxiety Scale (LSAS) is used to evaluate the intensity of fear and avoidance related to confrontation with social situations.
  The intensity of anxiety is rated separately from 0 (none) to 3 (severe) and the frequency of avoidance: 0 (never = 0%) to 3 (usual = 67 to 100%).
  We can use several different scores depending on the dimensions we are interested in (performance vs social interaction or anxiety vs. avoidance).
  The overall score is also widely used, it ranges from 0 to 144. The French norms are as follows: • 56-65: indicates a moderate social phobia;
  * 66-80: indicates a marked social phobia;
  * 81-95: indicates a severe social phobia; •> 95: indicates a very severe social phobia.
Yale-Brown Scale(Y-BOCS) | 3 months
  The rating scale is designed to rate the severity and type of symptoms in patients with obsessive compulsive disorder (OCD).
  The scale includes 10 items that measure 5 dimensions: duration, discomfort in daily life, anxiety, resistance, degree of control.
  Each item is rated from 0 (no symptoms) to 4 (extreme symptom). The scale makes it possible to distinguish an obsession score: addition of the 5 items (0 ≤ score ≤ 20) and a compulsion score: addition of the 5 items (0 ≤ score ≤ 20).
  According to the total score obtained (0 ≤ score ≤ 40), we will distinguish: • 10-18: light OCD causing distress but not necessarily dysfunction; the help of a third person is not claimed;
  * 18-25: distress and disability;
  * ≥ 30: severe disability requiring outside help.

CONTACTS AND LOCATIONS:
Overall Officials: SONIE SANDRINE, MD PH, Principal Investigator — Centre Hospitalier le Vinatier (BRON, France)
Locations (1):
- Centre hospitalier Le Vinatier, Bron, AURA, France

IPD SHARING:
Plan to Share IPD: No